CLINICAL TRIAL: NCT05571930
Title: Outcomes of Secondary Endovascular Aortic Repair After Initial Aortic Cross Replacement by a Frozen Elephant Trunk
Brief Title: Outcomes of Secondary Endovascular Aortic Repair After Initial Frozen Elephant Trunk Procedure
Status: Completed | Type: Observational
Sponsor: University Paul Sabatier of Toulouse (Other)
Collaborators: Jean Porterie, MD (Unknown); Thibaut Boisroux, MD (Unknown); Bertrand Marcheix, MD, PhD (Unknown); Jean Baptiste Ricco, MD, PhD (Unknown); Xavier Chaufour, MD, PhD (Unknown)
Responsible Party: Principal Investigator, Aurélien Hostalrich, Hostalrich Aurelien, MD, University Paul Sabatier of Toulouse
Other Study IDs: TEVAR after THX
Record Dates: First submitted 2022-05-24; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Thoraco-abdominal Aneurysm; Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Secondary TEVAR after initial FET procedure — Under general anesthesia, via percutaneous femoral access, the investigators implant a TEVAR in the endovascular part of a FET. This secondary connexion is indicated in case distal thoracic aortic involvement such as aneurysm or dissection.

SUMMARY:
Objective Complex aortic pathology has been revolutionized with the use of hybrid prostheses such as the Thoraflex® Hybrid Frozen Elephant Trunk (FET). The aim of this study was to evaluate the midterm results of secondary extension of the FET by thoracic endovascular aortic repair (TEVAR). Few data are present in the literature regarding the outcomes of this secondary treatment.

The investigators perform a prospective study between 2015 and 2022 in a tertiary aortic center on all consecutive patients having undergone TEVAR after FET implantation. The TEVAR endograft covered most of the 10 cm FET module with 2 to 4 mm oversizing. All patients were monitored by computerized angiography (CTA) at 6-month and yearly thereafter.

The aim of this study was the feasibility of theses secondary connexion and the mid term outcomes of the endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

Patient with aortic cross replacement by FET and

* Type 1 and Type 2 Thoracoabdominal aneurysm (TAAA) with a diameter at > 6 cm or
* an aortic dissection, Type A (TAAD) or Type B (TBAD) with either organ malperfusion due to compression of the true channel or aneurysmal evolution of the dissected aorta, or
* A defect in the expansion of the FET module

Exclusion Criteria:

* No aortic cross replacement by FET

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with aortic cross replacement by FET who are indicated for a secondary connexion in emergency :
  Aortic type A dissection with organ malperfusion Defect in the expansion of the FET module
  or in chronical evolution: Type 1 and Type 2 Thoracoabdominal aneurysm (TAAA) with a diameter at > 6 cm Aneurysmal evolution of the false lumen of a dissected aorta.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Absence of endoleak after secondary connexion | yearly thereafter up to 5 years
  Absence of Type 1A endoleak

SECONDARY OUTCOMES:
Feasibility of the secondary connexion | During the surgery
  Absence of failed procedure
Absence of endoleak after secondary connexion | early thereafter up to 5 years
  Absence of Type 3 endoleak

IPD SHARING:
Plan to Share IPD: No
Data are anonymised in our local prospective database shared between all investigators.